CLINICAL TRIAL: NCT04278339
Title: Study of Electrophysiological Markers Related to the Cognitive and Affective Processes Behind Empathic Behaviour in Schizophrenic Spectrum Disorder
Acronym: SchizoEmp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-PP-14
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROLLED SUBJECTS (Experimental): In this arm, only controlled subjects (pathological-free) will be investigated.
  Interventions: Other: Evoked Related Potentials
- PATIENTS (Experimental): In this arm, only patients with scyzophrenic syndrome will be investigated.
  Interventions: Other: Evoked Related Potentials

INTERVENTIONS:
Other: Evoked Related Potentials — Evoked Related Potentials are measured by means of electroencephalography. During this measure, 2 informatic task will be performed to evaluated evoked related potentials.

SUMMARY:
Disorders of social cognition, and empathy more specifically, are at the heart of schizophrenic pathology in that they are strongly linked to the social handicap of patients. It is therefore necessary to refine our knowledge of the cognitive and affective processes behind this empathic disorder and to identify objective and easily measurable markers (related to brain functioning collected by electroencephalography) of these processes with the subsequent aim of improving their management. It is also relevant to question the trait/status nature of these empathic disorders by studying these markers in individuals presenting more or less marked schizotypic traits and therefore more or less at risk of developing schizophrenia. Studying the possibility that empathy disorders may be part of the factors of developmental vulnerability for schizophrenia and identifying objective markers of this vulnerability could allow, in case of development of the pathology, a more rapid diagnosis and a more effective management.

ELIGIBILITY:
Inclusion Criteria:

* Common to all: good command of the French language, right-handed.
* Specific to patients: diagnosis of schizophrenia or schizoaffective disorder, clinical state stabilized according to the treating psychiatrist.

Exclusion Criteria:

* Common to all: having suffered a head injury with loss of consciousness lasting more than 5 minutes, participating in another project at the time of the present study, presenting an addiction to a toxic substance (excluding tobacco), presenting a mental retardation or neurological disorder (verified by a pre-recruitment interview and the administration of the Mini International Neuropsychiatric Interview for control subjects and on the basis of the information in the medical file for patients).
* Patient-specific: significant change (according to the doctor) in treatment in the previous month, currently hospitalized.
* Specific to controls: taking a psychoactive drug, having a mental disorder, being first-degree related to a patient with a disorder other than schizophrenia or schizoaffective disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evoked Related Potentials | On the first day
  Amplitude of modulations of the electrophysiological signal

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pasteur - Service de Psychiatrie, Nice, France

IPD SHARING:
Plan to Share IPD: No